CLINICAL TRIAL: NCT04670978
Title: Efficacy and Safety of Abraxane With Bevacizumab Biosimilar in Patients With Recurrent, Platinum-resistant Epithelial Ovarian Cancer：A Multi-center, Prospective, One-arm, Phase II Study
Brief Title: Abraxane With Bevacizumab Biosimilar in Patients With Recurrent, Platinum-resistant Epithelial Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Beihua Kong, Head of gynaecology and obstetrics, Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AB-PRR-EOC
Record Dates: First submitted 2020-12-05; First posted 2020-12-17 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Objective Response Rate
Keywords: epithelial ovarian cancer; platinum-resistant recurrent; Abraxane; Bevacizumab Biosimilar
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- albumin-bound paclitaxe combined with bevacizumab biosimilar (Experimental): albumin-bound paclitaxel, 260mg/m2，ivdrip，D1，once every three weeks bevacizumab biosimilar, 10mg/kg，ivdrip，D1, once every three weeks
  Interventions: Drug: albumin-bound paclitaxe combined with bevacizumab biosimilar

INTERVENTIONS:
Drug: albumin-bound paclitaxe combined with bevacizumab biosimilar — albumin-bound paclitaxe, 260mg/m2, every 3 weeks, 6cycles, bevacizumab biosimilar, 10mg/kg, every 3 weeks, continue until PD or unaccceptable toxicity

SUMMARY:
The study is a multi-center, prospective, one-arm, phase II clinical trial. It is tend to examine the safety and efficacy of combining abraxane(albumin-bound paclitaxel） and bevacizumab to treat patients with recurrent, platinum-resistant primary epithelial ovarian cancer, fallopian tube cancer or peritoneal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent or progressive primary EOC, fallopian tube carcinoma or peritoneal carcinoma (PC) within 6 months of their last previous platinum therapy
2. Patients had received at least one prior line of platinum-based chemotherapy
3. Patients were required to have one measurable disease for assessment according to RECIST version 1.1 or determined CA125 level according to GCIG
4. Eastern Cooperative Oncology Group (ECOG) Performance Status rating of 0-1
5. life expectancy ≥3 months
6. ≥30 days after surgery, the body has recovered and there is no active infection
7. Patients had received at least 1 prior line of platinum-based chemotherapy and were recurrent or progressed within 6 months after the end of the last platinum-based regimen
8. Must have adequate hematologic and hepatic function
9. Subjects of childbearing age must agree to use effective contraception during the trial period and negative for serum or urine pregnancy test
10. Patient provides voluntary written informed consent

Exclusion Criteria:

1. Previously received bevacizumab.
2. History of other invasive malignancy with the exception of nonmelanoma skin cancer
3. Participate in other drug trials
4. Blood pressure of >150/100 mmHg on antihypertensive medications
5. Previous history of hypertensive crisis or hypertensive encephalopathy
6. Diagnosed with unstable angina per NYHA or Grade 2 or greater congestive heart failure
7. The history of myocardial infarction within 6 months
8. The history of stroke or transient ischemic attack within 6 months of enrollment
9. Clinically significant vascular disease (e.g., aortic aneurysm, aortic dissection) or symptomatic peripheral vascular disease
10. Bleeding diathesis or coagulopathy
11. Presence of central nervous system or brain metastases
12. Pre-existing peripheral neuropathy of Grade ≥ 2
13. Major surgery was performed within 28 days prior to enrollment
14. Partial or complete ileus within 3 months prior to study enrollment
15. A biopsy or other minor surgery within 7 days prior to study enrollment
16. Positive pregnancy test or is lactating
17. Abdominal fistula, gastrointestinal perforation or abscess accumulation in the abdominal cavity within 6 months prior to study enrollment
18. Severe, nonhealing wound, ulcer, or bone fracture
19. Serious intercurrent medical or psychiatric illness, including serious active infection
20. Uncontrolled systemic infections require antiinfective treatment
21. Proteinuria at screening as demonstrated by either
22. Urine protein:creatinine (UPC) ratio ≥ 1.0 at screening OR
23. Urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible)
24. Known to be allergic, highly sensitive or intolerant to investigational drugs or their excipients

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
objective response rate | Assessed at the end of 6 cycle(each cycle is 21 days)
  Radiologic imaging was scheduled to be performed at baseline, after every third treatment cycle, and at the end of treatment or time of progression unless it was done in the previous four weeks. Response was evaluated using RECIST version 1.0 guidelines, where complete response (CR) is the disappearance of all target lesions; partial response (PR) is >=30% decrease in the sum of the longest diameter of target lesions; objective response rate (ORR) = CR+PR

SECONDARY OUTCOMES:
6-month progression-free survival rate | assessed up to 6 months
  the percentage of participants with no progression event at 6 months after starting study treatment
progression-free survival | up to 3 years
  PFS was measured from day 1 of treatment until time of progression (assessed every 12 weeks) or death, whichever came first
overall survival | assessed up to 3 years
  Overall survival is defined as the time from treatment start until death from any cause
Disease control rate | Assessed at the end of 6 cycle(each cycle is 21 days)
  the percentage of complete and partial response as well as stable disease

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No